CLINICAL TRIAL: NCT00654875
Title: A 10 Week, Randomized, Double-blind, Parallel Group, Multi-center Study to Evaluate the Efficacy and Safety of Once Daily Dosing of Aliskiren (300 mg qd) to Twice Daily Dosing of Aliskiren (150 mg Bid) in Patients With Essential Hypertension.
Brief Title: Efficacy and Safety of Once Daily Dosing of Aliskiren (300 mg (qd) Once a Day) to Twice Daily Dosing of Aliskiren (150 mg (Bid) Twice a Day) in Treating Moderate Hypertension.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2403
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren 300 mg (Once a Day) (Experimental): Participants received Aliskiren 300 mg tablet + Placebo to Aliskiren matching 150 mg tablet daily in the morning and Placebo to Aliskiren matching 150 mg tablet daily in the evening for a total of 10 weeks.
  Interventions: Drug: Aliskiren; Drug: Placebo to Aliskiren
- Aliskiren 150 mg (Twice a Day) (Experimental): Participants received Aliskiren 150 mg tablet + Placebo to Aliskiren matching 300 mg tablet daily in the morning and Aliskiren 150 mg tablet daily in the evening for the first 6 weeks then for the next 4 weeks received Aliskiren 300 mg tablet + Placebo to Aliskiren matching 150 mg tablet daily in the morning and Placebo to Aliskiren matching 150 mg tablet daily in the evening.
  Interventions: Drug: Aliskiren; Drug: Placebo to Aliskiren

INTERVENTIONS:
Drug: Aliskiren — Aliskiren supplied in 150 mg and 300 mg tablets.
  Other Names: Tekturna, Rasilez
Drug: Placebo to Aliskiren — Placebo to Aliskiren matching 150 and 300 mg tablets

SUMMARY:
This study will compare the safety and efficacy of once daily dosing of aliskiren to twice daily dosing of aliskiren in patients with moderate hypertension

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of uncomplicated essential hypertension; newly diagnosed or who have not received antihypertension medication within 4 weeks of visit 1 must have an office cuff mean sitting Diastolic Blood pressure (msDBP) > 100 mmHg and < 110 mmHg at visit 1. If patient is receiving antihypertensive treatment, must have a cuff msDBP > 95 mmHg and < 110 mmHg at visit 1
* Prior to randomization, all patients must have an office cuff msDBP >or= 100 mmHg and <or = 110 mmHg.

Exclusion Criteria:

* Participation in another aliskiren trial or previous treatment with aliskiren during last 6 months and who qualified to be randomized or enrolled into the active drug treatment period
* Pregnant or nursing women
* Women of child bearing potential unwilling to use protocol specific contraceptive methods
* Office cuff blood pressure of msDBP ≥ 112 mmHg and/or mean sitting Systolic Blood Pressure (msSBP) ≥ 200 mmHg).
* Secondary form of hypertension
* History of heart failure New York Heart Association (NYHA Class II, III and IV)
* Previous history of hypertensive encephalopathy or stroke, transient ischemic attack (TIA), heart attack, coronary bypass surgery or any percutaneous coronary intervention (PCI)
* Elevated Serum potassium (> or = 5.3 mEq/L (mmol/L) at Visit 1
* Type 1 or Type 2 diabetes mellitus not well controlled
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis
Locations (3):
- Investigative Site, Zanesville, Ohio, United States
- Investigative Site, Frankfurt, Germany
- Investigative Site, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Started | 164 | 164
Completed | 147 | 147
Not Completed | 17 | 17
Not completed — Adverse Event | 5 | 5
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Protocol Violation | 3 | 3
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Abnormal Test Procedure Result(s) | 1 | 0
Not completed — Administrative Problems | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day) | Total
Number analyzed (Participants) | 164 | 164 | 328
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (10.3) | 54 (10.2) | 54 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 77 | 140
  Male | 101 | 87 | 188

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the Mean 24-hour Ambulatory Diastolic Blood Pressure (MADBP)
Description: An Ambulatory Blood Pressure Monitoring (ABPM) device was attached to the non-dominant arm of the participant. The mean of Blood Pressure readings during the 24 hour period were calculated. The difference of the 24 hour MADBP from baseline to the 24 hour MADBP at 6 weeks was calculated using an Analysis of covariance (ANCOVA) model with baseline mean 24 hour ambulatory diastolic blood pressure as a covariate.
Time Frame: Baseline, Week 6
Population: Participants from the Full analysis set (consisting of all randomized patients) for whom data was available at Baseline and Week 6.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 139 | 127
mm Hg | -4.10 (0.60) | -5.24 (0.64)

2. Secondary Outcome: Change From Baseline to Week 6 in the Mean Ambulatory Diastolic Blood Pressure (MADBP) During the Last 3 Hours of the 24-hour Dosing Period
Description: An Ambulatory Blood Pressure Monitoring (ABPM) device was attached to the non-dominant arm of the participant. The mean of Blood Pressure readings during the 22-24 hour period were calculated. The difference from the last 3 hours MADBP at baseline to the last 3 hour MADBP at Week 6 was calculated using an ANCOVA model with baseline mean 24 hour ambulatory diastolic blood pressure as a covariate.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 136 | 121
mm Hg | -5.03 (0.77) | -5.24 (0.81)

3. Secondary Outcome: Change From Baseline to Week 6 in the Mean Ambulatory Systolic Blood Pressure (MASBP) During the Last Three Hours of the 24-hour Dosing Period
Description: An Ambulatory Blood Pressure Monitoring (ABPM) device was attached to the non-dominant arm of the participant. The mean of Blood Pressure readings during the 22-24 hour period were calculated. The difference from the last 3 hours MASBP at baseline to the last 3 hour MASBP at Week 6 was calculated using an ANCOVA model with baseline mean 24 hour ambulatory systolic blood pressure as a covariate.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 136 | 121
mm Hg | -6.39 (1.04) | -7.12 (1.10)

4. Secondary Outcome: Change From Baseline to Week 6 in the Mean 24-hour Ambulatory Systolic Blood Pressure (MASBP)
Description: An Ambulatory Blood Pressure Monitoring (ABPM) device was attached to the non-dominant arm of the participant. The mean of Blood Pressure readings during the 24 hour period were calculated. The difference of the 24 hour MASBP from baseline to the 24 hour MASBP at 6 weeks was calculated using an ANCOVA model with baseline mean 24 hour ambulatory systolic blood pressure as a covariate.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 139 | 127
mm Hg | -5.74 (0.87) | -7.44 (0.92)

5. Secondary Outcome: Change From Baseline to Week 6 in the Mean Sitting Systolic and Mean Sitting Diastolic Blood Pressure
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using a calibrated standard sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1-2 minute intervals and the mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure for that visit. A negative number indicates lowered blood pressure. The ANCOVA model used baseline as a covariate.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 158 | 156
mm Hg
  Diastolic Blood Pressure | -10.30 (0.66) | -10.57 (0.67)
  Systolic Blood Pressure | -11.72 (1.11) | -13.10 (1.11)

6. Secondary Outcome: Percentage of Participants Achieving Blood Pressure Control at Week 6
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using a calibrated standard sphygmomanometer. The mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure at visit 3 (week 6).
  Blood pressure control was defined as having a mean sitting diastolic blood pressure (msDBP) <90 mm Hg and a mean sitting systolic blood pressure (msSBP) <140 mm Hg.
Time Frame: Week 6
Population: Participants from the Full analysis set (consisting of all randomized patients) for whom data was available at Week 6.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 158 | 156
Percentage of participants | 24.7 | 26.9

7. Secondary Outcome: Percentage of Participants Achieving Blood Pressure Control at the End of the Study (Week 10)
Description: After the patient had been sitting for 5 minutes, with the back supported and both feet placed on the floor, systolic and diastolic blood pressures were measured 3 times using a calibrated standard sphygmomanometer. The mean of these 3 sitting blood pressure measurements was used as the average sitting blood pressure at visit 4 (week 10).
  Blood pressure control was defined as having a mean sitting diastolic blood pressure (msDBP) <90 mm Hg and a mean sitting systolic blood pressure (msSBP) <140 mm Hg.
Time Frame: Week 10
Population: Participants from the Full analysis set (consisting of all randomized patients) for whom data was available at Week 10.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Number analyzed (Participants) | 154 | 155
Percentage of participants | 24.0 | 27.7

ADVERSE EVENTS:
Time Frame: 10 Weeks
Arm/Group | Aliskiren 300 mg (Once a Day) | Aliskiren 150 mg (Twice a Day)
Serious Adverse Events (participants affected / at risk) | 2/164 | 2/164
Other Adverse Events (participants affected / at risk) | 0/164 | 0/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 300 mg (Once a Day) (N=164) | Aliskiren 150 mg (Twice a Day) (N=164)
Appendicitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.